CLINICAL TRIAL: NCT04993521
Title: Ultrasound Guided Bilateral Superficial Cervical Plexus Block Versus Local Wound Infiltration in Patients Undergoing Total Thyroidectomy: A Randomized Controlled Study
Brief Title: Ultrasound Guided Bilateral Superficial Cervical Plexus Block in Patients Undergoing Total Thyroidectomy.
Acronym: BSCPB_Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Linkoeping (Other)
Collaborators: Ahmed Mohamed Abdelrahman (Unknown); Mahmoud Ahmed Mewafy (Unknown); Abdelrhman Alshawadfy (Unknown); Haidi Abd-Elzaher (Unknown); Hamada Fathy (Unknown); Mohamed Faisal (Unknown)
Responsible Party: Principal Investigator, Folke Sjoberg, professor, University Hospital, Linkoeping
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BSCPB_Block
Record Dates: First submitted 2021-06-10; First posted 2021-08-06 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-07

CONDITIONS: Analgesia Obtained With a Local Wound Infiltration of Lidocain; Analgesia Obtained With a Ultrasound Guided Cervical Plexus Block Using Lidocain; Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: A Randomized Controlled Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- bilateral superficial cervical plexus block (BSCPB) (Active Comparator): Analgesia obtained by a ultrasound guided cervical plexus block using lidocain
  Interventions: Procedure: Block type
- local wound infiltration (LWI) (Active Comparator): Analgesia obtained by local wound infiltration of lidocain
  Interventions: Procedure: Block type

INTERVENTIONS:
Procedure: Block type — Regular block type
  Other Names: Ultrasound guided bilateral superficial cervical plexus nerve block

SUMMARY:
The present study compared the efficacy of bilateral superficial cervical plexus block (BSCPB) versus local wound infiltration (LWI) regarding the postoperative opioid consumption in patients undergoing total thyroidectomy

DETAILED DESCRIPTION:
We performed a double-blind, randomised, controlled trial that recruited patients undergoing total thyroidectomy at the Suez Canal University Hospital during the period between February 2019 and January 2021. Patients were eligible if they were older than 20 years, had an American Association of Anesthesiologists' (ASA) level of I-II, and were scheduled for total thyroidectomy. We excluded patients with documented allergies to the study's intervention materials, moderate-to-severe obesity, > 1st-degree heart block, chronic pulmonary or cardiac diseases, hepatic or renal dysfunction, and/or coagulopathies. All patients were required to fill out informed consent before enrollment.

Eligible patients were randomly allocated in a 1:1 ratio to receive BSCPB or LWI using the computer software program (www. Randmizer.org) and allocation sequences were done using opaque, closed envelopes. The BSCPB group received BSCBP (after general anaesthesia but before the start of surgery) from two syringes containing ropivacaine 0.5 % and LWI with saline. The LWI group received LWI with ropivacaine 0.5% and the BSCPB from two syringes containing saline.

The primary outcome of the present study was postoperative opioid consumption in the first postoperative day. The secondary outcomes included the total intraoperative fentanyl and isoflurane consumption, time to first required analgesic, and VAS during the first 24 hours postoperatively.

ELIGIBILITY:
Inclusion Criteria:

ASA I-II, and were scheduled for total thyroidectomy

-

Exclusion Criteria:

documented allergy to study's intervention, moderate-to-severe obesity, > 1st-degree heart block, chronic pulmonary or cardiac diseases, hepatic or renal dysfunction, and/or coagulopathies.

All patients were required to fill the informed consent before enrollment.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-05-15 (Actual)

PRIMARY OUTCOMES:
postoperative opioid consumption in the first postoperative day | 24 hours
  postoperative opioid consumption in the first postoperative day in milligrams

SECONDARY OUTCOMES:
total intraoperative fentanyl (mg) and isoflurane consumption (ml) | 6 hours
  total intraoperative fentanyl and isoflurane consumption in micrograms and ml
time to first required analgesic | 6 hours
  time to first required analgesic
VAS (10 cm; range): Pain average (VAS) for the first 24 hours postoperatively | every 6 hours until 24 hours postoperatively
  VAS (10 cm; range) Pain average (VAS) for the first 24 hours postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Linköping University Hospital, Linköping, Sweden

IPD SHARING:
Plan to Share IPD: No
Can be shared on reasonable terms